CLINICAL TRIAL: NCT01161862
Title: Integration of Continuous Glucose Monitoring Into a Bi-Hormonal Closed-Loop Artificial Pancreas for Automated Management of Type 1 Diabetes
Brief Title: Integration of Continuous Glucose Monitoring Into a BiHormonal Closed-Loop Artificial Pancreas
Acronym: CL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Massachusetts General Hospital (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Juvenile Diabetes Research Foundation (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Edward R. Damiano, Associate Professor of Biomedical Engineering, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-29293; 1R01DK085633-01 (NIH)
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus
Keywords: Closed-loop; Artificial pancreas; Bi-hormonal; Insulin; Glucagon; Diabetes mellitus type 1
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bi-hormonal with meal-priming bolus (Experimental): The first meal-priming bolus was solely based on weight (0.05 U/kg), after which meal-priming boluses were automatically adapted by the control system online targeting 75% of the anticipated insulin needed in the first four hours after the start of the meal
  Interventions: Device: Bi-hormonal (insulin and glucagon) artificial pancreas
- Bi-hormonal without meal-priming bolus (Experimental): The insulin controller was entirely reactive to CGMG; there were no meal priming boluses and no meal announcements
  Interventions: Device: Bi-hormonal (insulin and glucagon) artificial pancreas

INTERVENTIONS:
Device: Bi-hormonal (insulin and glucagon) artificial pancreas — Subjects wore a bionic pancreas consisting of a continuous glucose monitor, an insulin pump and a glucagon pump

SUMMARY:
The investigators hypothesize that our closed-loop glucose-control system can provide BG control in subjects with type 1 diabetes using the estimated BG signal from a CGM as the input signal to the controller.

DETAILED DESCRIPTION:
To test the safety and efficacy of our control system in the bi-hormonal configuration in regulating BG in adults (18 years of age or older) and in children (12-17 years of age) with type 1 diabetes based on interstitial-fluid (ISF) glucose data from a CGM. Experiments will be 51 hours in length incorporating 6 meals and two (night) sleep periods. In order to evaluate the effect of exercise on BG control, the last 48 hours of the experiment will be divided into two 24 hour blocks, the second of which will contain a period of structured exercise near the beginning of the block.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 years or older with clinical type 1 diabetes for at least one year
* Weight > 41 kg
* Otherwise healthy (mild chronic disease allowed if well controlled)
* Diabetes managed using an insulin infusion pump and rapid- or very-rapid-acting insulins
* Body mass index (BMI) between 20 and 35 for subjects >18 years of age or BMI between the 5th and 95th percentile for age for subjects < 18 years of age
* Total daily dose (TDD) of insulin that is < 1 U/kg
* Stimulated C-peptide < 0.1 nmol/L at 90 minutes after liquid mixed meal by DCCT protocol
* Hemoglobin A1c <= 9%
* Prescription medication regimen stable for 1 month

Exclusion Criteria:

* Unable to provide informed consent for subjects > 18 years of age or unable to provide assent if < 18 years of age
* Unable to comply with study procedures
* Current participation in another diabetes-related clinical trial other than one that is primarily observational in nature. Potential subjects enrolled in trials of passive monitoring equipment are not excluded.
* Anemia (HCT less than normal for age and sex)
* Alanine aminotransferase > 3 fold above upper limit of normal
* Untreated or inadequately treated hyperthyroidism or hypothyroidism
* Pregnancy
* Renal insufficiency (creatinine clearance ≤ 50 ml/min)
* Any known history of coronary artery disease
* Abnormal EKG including, but not limited to evidence of active ischemia, prior myocardial infarction, proximal LAD critical stenosis (Wellen's sign), arrhythmia, tachycardia, and prolonged QT interval (> 440 ms)
* Congestive heart failure
* History of TIA or stroke
* Acute illness or exacerbation of chronic illness
* History of seizures
* History of pheochromocytoma (fractionated metanephrines will be tested in patients with history suggestive of pheochromocytoma)
* History of adrenal disease or tumor
* History of pancreatic tumor, including insulinoma
* History of impaired gastric motility or gastroparesis requiring pharmacological or surgical treatment
* Current alcohol abuse (intake averaging > 3 drinks daily in last 30 days) or substance abuse (any use within the last 6 months of controlled substances without a prescription)
* Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year)
* Impaired cognition or altered mental status.
* Hypertension (blood pressure > 140/90 or > 95% for age, height and weight in subjects < 18 years of age) at the time of screening
* Use of medications that reduce gastric motility (e.g. narcotics, anti-spasmodics, anticholinergics).
* Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference
* Use non-insulin, injectable anti-diabetic medications
* History of adverse reaction to glucagon (including allergy) besides nausea and vomiting.
* Established history of latex, adhesive, or tape allergy
* Inadequate venous access
* History of allergy to aspirin or any history of aspirin intolerance, including Reye syndrome, or gastric ulcer or bleeding associated with salicylates
* Blood dyscrasia or bleeding diathesis, such as hemophilia, Von Willebrands disorder, and idiopathic thrombocytopenic purpura (ITP)
* Peptic ulcer
* Unable to perform 30 minutes of moderate exercise on a treadmill or exercise bicycle
* Unable or unwilling to discontinue dietary supplements for at least 2 weeks prior to each CRC admission
* History of celiac disease

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Damiano ER, El-Khatib FH, Zheng H, Nathan DM, Russell SJ. A comparative effectiveness analysis of three continuous glucose monitors. Diabetes Care. 2013 Feb;36(2):251-9. doi: 10.2337/dc12-0070. Epub 2012 Dec 28. PMID 23275350
- [Derived] Russell SJ, El-Khatib FH, Nathan DM, Magyar KL, Jiang J, Damiano ER. Blood glucose control in type 1 diabetes with a bihormonal bionic endocrine pancreas. Diabetes Care. 2012 Nov;35(11):2148-55. doi: 10.2337/dc12-0071. Epub 2012 Aug 24. PMID 22923666
- See also: Related Info — http://www.artificialpancreas.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve adult and twelve pediatric subjects with type 1 diabetes and no endogenous insulin secretion participated in two 51-h experiments. The protocol was approved by the Massachusetts General Hospital (MGH) and Boston University Human Research Committees
Groups:
- Bi-hormonal Bionic Pancreas With Meal-priming Bolus: The first meal-priming bolus was solely based on weight (0.05 U/kg), after which meal-priming boluses were automatically adapted by the control system online targeting 75% of the anticipated insulin needed in the first four hours after the start of the meal.
- Bi-hormonal Bionic Pancreas With no Meal-priming Bolus: Bi-hormonal bionic pancreas with no meal-priming bolus. The controller was entirely reactive to CGMG; there were no meal priming boluses and no meal announcements
Period: Overall Study
Arm/Group | Bi-hormonal Bionic Pancreas With Meal-priming Bolus | Bi-hormonal Bionic Pancreas With no Meal-priming Bolus
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bi-hormonal Pancreas With Meal-priming Bolus: An automatically adapting meal priming bolus was given by the controller at the time each meal was presented
- Bi-hormonal Pancreas Without Meal-priming Bolus: The insulin controller was entirely reactive to CGMG; there were no meal priming boluses and no meal announcements
- Total: Total of all reporting groups
Arm/Group | Bi-hormonal Pancreas With Meal-priming Bolus | Bi-hormonal Pancreas Without Meal-priming Bolus | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 12
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (17.7) | 30.5 (19.0) | 30 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Plasma Blood Glucose Achieved by the Bionic Pancreas (mg/dl)
Time Frame: 48 hours
Population: Overall number of participants was 24, 12 in each arm
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Bionic Pancreas With Automated Meal-priming Bolus: Bi-hormonal bionic pancreas
  Bi-hormonal (insulin and glucagon) artificial pancreas
Arm/Group | Bionic Pancreas With Automated Meal-priming Bolus | Bionic Pancreas Without Automated Meal-priming Bolus
Number analyzed (Participants) | 12 | 12
mg/dl
  Adults: number analyzed (Participants) | 6 | 6
  Adults | 132 (3) | 146 (9)
  Adolescents: number analyzed (Participants) | 6 | 6
  Adolescents | 162 (6) | 175 (9)

2. Secondary Outcome: Percentage of Time Spent With Blood Glucose < 60 mg/dl
Time Frame: 48 hours
Population: Overall number of participants=24 (12 in each arm)
Measure: Mean (Standard Deviation); unit: percentage of total time
Arm/Group | Bionic Pancreas With Automated Meal-priming Bolus | Bionic Pancreas Without Automated Meal-priming Bolus
Number analyzed (Participants) | 12 | 12
percentage of total time
  Adults: number analyzed (Participants) | 6 | 6
  Adults | 2.3 (3.9) | 1.4 (2.7)
  Adolescents: number analyzed (Participants) | 6 | 6
  Adolescents | 0.1 (0.2) | 0.1 (0.2)

3. Secondary Outcome: Percentage of Time Spent With Blood Glucose <70 mg/dl
Time Frame: 48 hours
Population: Overall number of participants=24 (12 in each arm)
Measure: Mean (Standard Deviation); unit: percentage of total time
Arm/Group | Bionic Pancreas With Automated Meal-priming Bolus | Bionic Pancreas Without Automated Meal-priming Bolus
Number analyzed (Participants) | 12 | 12
percentage of total time
  Adults: number analyzed (Participants) | 6 | 6
  Adults | 5.1 (6.7) | 3.6 (4.5)
  Adolescents: number analyzed (Participants) | 6 | 6
  Adolescents | 0.3 (0.5) | 0.4 (0.7)

4. Secondary Outcome: Percentage of Time Spent With Blood Glucose 70-180 mg/dl
Time Frame: 48 hours
Population: Overall number of participants=24 (12 in each arm)
Measure: Mean (Standard Deviation); unit: percentage of total time
Arm/Group | Bionic Pancreas With Automated Meal-priming Bolus | Bionic Pancreas Without Automated Meal-priming Bolus
Number analyzed (Participants) | 12 | 12
percentage of total time
  Adults: number analyzed (Participants) | 6 | 6
  Adults | 80 (6) | 70 (9)
  Adolescents: number analyzed (Participants) | 6 | 6
  Adolescents | 68 (8) | 60 (4)

5. Secondary Outcome: Insulin Total Daily Dose
Time Frame: 48 hours
Population: Overall number of participants=24 (12 in each arm)
Measure: Mean (Standard Deviation); unit: u/kg/day
Arm/Group | Bionic Pancreas With Automated Meal-priming Bolus | Bionic Pancreas Without Automated Meal-priming Bolus
Number analyzed (Participants) | 12 | 12
u/kg/day
  Adults: number analyzed (Participants) | 6 | 6
  Adults | 0.6 (0.2) | 0.7 (0.2)
  Adolescents: number analyzed (Participants) | 6 | 6
  Adolescents | 1.1 (0.2) | 1.2 (0.2)

6. Secondary Outcome: Number of Carbohydrate Interventions for Hypoglycemia
Time Frame: 48 hours
Population: Overall number of participants=24 (12 in each arm)
Measure: Number; unit: Carbohydrate Interventions
Groups:
- Bi-hormonal With Meal Priming Bolus: Bi-hormonal bionic pancreas
  Bi-hormonal (insulin and glucagon) artificial pancreas
Arm/Group | Bi-hormonal With Meal Priming Bolus | Bi-hormonal Without Meal Priming Bolus
Number analyzed (Participants) | 12 | 12
Carbohydrate Interventions | 12 | 10

7. Secondary Outcome: Number of Blood Glucose Events < 70 mg/dl
Time Frame: 48 hours
Measure: Number; unit: Number of events
Arm/Group | Bi-hormonal With Meal Priming Bolus | Bi-hormonal Without Meal Priming Bolus
Number analyzed (Participants) | 12 | 12
Number of events | 59 | 48

8. Secondary Outcome: Nadir Blood Glucose in Each Arm
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Bionic Pancreas Without Automated Meal-priming Bolus: Bi-hormonal bionic pancreas
  Bi-hormonal (insulin and glucagon) artificial pancreas
Arm/Group | Bionic Pancreas With Automated Meal-priming Bolus | Bionic Pancreas Without Automated Meal-priming Bolus
Number analyzed (Participants) | 12 | 12
mg/dl | 65.9 (17.4) | 66.4 (17.8)

ADVERSE EVENTS:
Time Frame: 51 hours per experiment
Groups:
- Bi-hormonal With Meal Priming Bolus: Bi-hormonal with adaptive meal priming bolus
- Bi-hormonal Without Meal Priming Bolus: Bi-hormonal with no meal announcements or meal priming boluses
Arm/Group | Bi-hormonal With Meal Priming Bolus | Bi-hormonal Without Meal Priming Bolus
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bi-hormonal With Meal Priming Bolus (N=12) | Bi-hormonal Without Meal Priming Bolus (N=12)
Nausea (General disorders) | 1 (1) | 1 (1) — The subject with the slowest insulin absorption and who received the most glucagon reported nausea on several occasions. However, the timing of these symptoms did not correspond to periods of high plasma glucagon levels

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No